CLINICAL TRIAL: NCT05651724
Title: Global Research Initiative for Patients Screening on MASH - Implementation of an International Transmural Patient Care Pathway
Brief Title: Global Research Initiative for Patients Screening on MASH
Acronym: GRIPonMASH
Status: Recruiting | Type: Observational
Sponsor: Julius Clinical (Industry)
Collaborators: UMC Utrecht (Other); Echosens (Industry); MIMETAS BV (Unknown); Nordic Bioscience A/S (Industry); Elevate BV (Unknown); Leiden University (Other); Amsterdam University Medical Center (Other); Andaluz Health Service (Other Government); National Research Council, Institute of Clinical Physiology, Italy (Other); Leiden University Medical Center (Other); Université Libre de Bruxelles (Other); University Hospital, Antwerp (Other); Catholic University of the Sacred Heart (Other); Medical Education Research And Innovation Center S.R.L. (Unknown); EUROPEAN LIVER PATIENTS ASSOCIATION (Unknown); Harokopio University (Other); General University Hospital, Prague (Other); Novo Nordisk A/S (Industry); Maastricht University (Other); Mercodia Aktiebolag (Unknown); EXIT071 BV (Unknown); European Atherosclerosis Society (Other); MetaDeq Limited (Unknown); Associação para Investigação e Desenvolvimento da Faculdade de Medicina (Unknown); Institute of Cardiometabolism and Nutrition, France (Other); University Hospital, Saarland (Other); Roche Pharma AG (Industry); Inventiva Pharma (Industry); Biocellvia (Unknown); Franciscus Gasthuis & Vlietland (Hospital) (Other)
Responsible Party: Sponsor
Other Study IDs: GOM
Record Dates: First submitted 2022-10-18; First posted 2022-12-15 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: MASH; MASLD; MASH With Fibrosis; Fibrosis, Liver; Steatosis of Liver; Type 2 Diabetes; Obesity; Metabolic Syndrome; Arterial Hypertension
Keywords: MASLD; MASH; Screening; Patient care pathway
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Diabetes Mellitus, Type 2; Obesity; Metabolic Syndrome; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood (plasma, serum, whole blood, DNA), liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
GRIPonMASH will assist (primary) health care providers clinicians to implement the latest patient care pathway, as described by the European Association for the Study of the Liver (EASL), to identify patients at risk of severe metabolic dysfunction-associated steatotic liver disease (MASLD) and to raise awareness. The primary objective is to implement a transmural patient care pathway, in order to identify patients with MASLD and its progressive form metabolic dysfunction-associated steatohepatitis (MASH) in primary care centres and clinics in 10 European countries.

DETAILED DESCRIPTION:
GRIPonMASH is an observational study in which 10.000 high risk patients (type 2 diabetes mellitus, metabolic syndrome, obesity or arterial hypertension) in 10 different European countries will be screened for the presence of MASLD, liver fibrosis and (at-rsik) MASH using at least two non-invasive tests (FIB-4 and FibroScan). Additional published and exploratory non-invasive test will also be investigated. Blood samples and liver biopsy material will be collected. Genomic, proteomic, metabolomic, lipidomic and fluxomic studies will be applied to gain a better understanding of the pathophysiology of MASLD and to identify (bio)markers that will help to detect patients at-risk. The predictive value of FIB-4 in relation to FibroScan results and liver biopsy will be analysed. Long-term follow-up of 5 years in all participants will provide insight into the natural history of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed subjects should fulfil criteria for diagnosis of type 2 diabetes mellitus or metabolic syndrome or obesity or arterial hypertension, following the study definitions.
* Subjects that are currently being treated for type 2 diabetes mellitus or metabolic syndrome or obesity or arterial hypertension, should have had a prior diagnosis based on study definitions.

Study definitions:

Type 2 diabetes mellitus

* At least 2 times a fasting glucose > 7,0 mmol/L
* Or elevated non-fasting glucose >11,1 mmol/L 2 hrs after OGTT
* Or HbA1c ≥48 mmol/mol (≥6.5%)
* Or being actively treated for previously diagnosed type 2 diabetes by a health care provider

Obesity

* Body mass index (BMI) > 30
* Or waist circumferences Caucasian: male ≥ 94 cm, female ≥ 80 cm South-Asian/Chinese: male ≥90 cm, female ≥80 cm Japanese: male ≥85 cm, female ≥90 cm

Arterial hypertension

* Systolic BP ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg
* Or being actively treated for previously diagnosed arterial hypertension by a health care provider

Metabolic syndrome

- Central obesity defined as waist circumference (see above), if BMI is >30 kg/m2, central obesity can be assumed and waist circumference does not need to be measured

AND any two of the following:

* Raised triglycerides: ≥ 150 mg/dL (1.7 mmol/L), or specific treatment for this lipid abnormality
* Reduced HDL cholesterol: < 40 mg/dL (1.03 mmol/L) in males, < 50 mg/dL (1.29 mmol/L) in females, or specific treatment for this lipid abnormality
* Raised blood pressure (BP): systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg, or treatment of previously diagnosed hypertension
* Raised fasting plasma glucose (FPG): FGP ≥ 100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes (if above >5.6 mmol/L or 100 mg/dL, an oral glucose tolerance test is strongly recommended, but is not necessary to define presence of the syndrome)

Exclusion Criteria:

* The patient is known with hepatitis B, C or HIV or any other liver condition (like hemochromatosis, sarcoidosis, Wilson's disease etc);
* The patient is known with any other condition that may lead to liver fibrosis or cirrhosis;
* The patient engages in (excessive) alcohol use: > 3 units/day in males [30 grams/day] and > 2 units/day in females [20 grams/day];
* The patient has a history or evidence of any other clinically significant condition or planned or expected procedure that in the opinion of the Investigator, may compromise the patient's safety or ability to be included in this study;
* The patient is an employee or contractor of the facility that is conducting the study or is a family member of the Investigator, sub-Investigator, or any Sponsor personnel;
* The patient is not able to understand the details of the protocol and/or is not able to provide written informed consent;
* The patient is pregnant or breastfeeding.
* The patient underwent bariatric surgery in the last 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged 18-75 years with a current or prior diagnosis of at least one of the following four conditions: type 2 diabetes mellitus or metabolic syndrome or obesity or arterial hypertension. Subjects who meet the inclusion and exclusion criteria will be enrolled at primary care centers in one of the 10 countries.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of liver steatosis and MASLD estimated by FibroScan CAP in patients at risk | Baseline
  Steatosis grade deduced from controlled attenuation parameter (CAP) measurement with Fibroscan
Prevalence of liver fibrosis estimated by FibroScan LSM in patients at risk | Baseline
  Fibrosis stage deduced from liver stiffness measurement (LSM) by vibration controlled transient elastography (VCTE) measurement with Fibroscan
Prevalence of at-risk MASH estimated by FAST score in patients at risk | Baseline
  At-risk MASH deduced from FAST score
*Subset of patients: prevalence of MASH in patients at risk | 16 or 30 weeks
  MASH diagnosis confirmed by histology (NAS/SAF criteria) upon liver biopsy; only in patients with >12 kPa at 1st FibroScan or >=8 kPa at 2nd FibroScan
Comparison of the prevalence of MASLD, liver fibrosis and (at-risk) MASH between the participating countries | Baseline (1-3) to 16/30 weeks for biopsy-confirmed MASH (4)
  Prevalence (see outcome 1-4) stratified per country
Evaluate added value of a 2-step pathway as compared to FibroScan only for detection of high-risk patients | Baseline
  Number of patients at risk identified by FIB-4 compared to numbers found using LSM by VCTE with FibroScan measurements, and numbers found in combination

SECONDARY OUTCOMES:
Build diagnostic model to identify MASH patients in a high-risk population | Baseline
  Possible model parameters are all baseline clinical characteristics reported in the eCRF
Genotypes related to MASH in different European countries: Exploratory | Baseline
  Genomic (GWAS) and proteomic analysis on collected blood samples
(Non-invasive) metabolite biomarkers identifying MASH in patients at risk: Exploratory | Baseline
  Mass-spectrometry (MS) based metabolomic and lipidomic analyses on collected blood and samples, both targeted and untargeted approaches.
Prevalence of co-morbidities and associated therapies (especially for CVD) in patients with MASH compared to those without, in high-risk patient populations | Baseline
  Prevalence of comorbidities, medication use, medical history
Identify prognostic factors/biomarkers for complications in patients with MASLD and MASH by 5 years follow up | Throughout follow-up (at 3 and 5 years)
  Disease progression and liver-related and non-liver related complications
Patient Reported Outcomes: Dietary habits and lifestyle | Baseline + throughout follow-up (at 3 and 5 years)
  14 item Mediterranean Diet Score; lifestyle surveys
*Subset of patients: Second FibroScan examination | 14 weeks
  CAP and LSM by VCTE at 2nd FibroScan examination
Longitudinal changes in liver assessments | Baseline, 14 weeks + throughout follow-up (at 3 and 5 years)
  Repeated CAP, LSM by VCTE and FAST measurements over time

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Castro Cabezas, MD/PhD, Principal Investigator — Sint Franciscus Gasthuis; Diederick E. Grobbee, MD/PhD/FESC, Principal Investigator — UMC Utrecht; Oscar H. Franco, MD/PhD/FESC/FFPH, Study Chair — UMC Utrecht
Locations (13):
- Belgium (2):
  - Hôpital Erasme, Cliniques Universitaires De Bruxelles, Brussels, Vlaams-brabant
  - Antwerp University Hospital, Antwerp
- 4th internal clinic General University Hospital, Prague, Bohemia, Czechia
- Hôpital de la Pitié Salpêtrière, Paris, Il-de-France, France
- Germany (2):
  - Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
- Harokopio University of Athens, Athens, Greece
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS (FPG), Università Cattolica del Sacro Cuore (UCSC), Rome, Lazio, Italy
- Netherlands (2):
  - Amsterdam UMC, Amsterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Rotterdam, South Holland
- ULSSM - Unidade Local de Saúde Santa Maria, E.P.E, Lisbon, Portugal
- Sacele Municipal Hospital, Săcele, Brașov County, Romania
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Jong VD, Alings M, Bruha R, Cortez-Pinto H, Dedoussis GV, Doukas M, Francque S, Fournier-Poizat C, Gastaldelli A, Hankemeier T, Holleboom AG, Miele L, Moreno C, Muris JWM, Ratziu V, Romero-Gomez M, Schattenberg JM, Serfaty L, Stefan DC, Tushuizen ME, Verheij J, Willemse J, Franco OH, Grobbee DE, Castro Cabezas M; GRIPonMASH consortium. Global research initiative for patient screening on MASH (GRIPonMASH) protocol: rationale and design of a prospective multicentre study. BMJ Open. 2025 May 30;15(5):e092731. doi: 10.1136/bmjopen-2024-092731. PMID 40447415
- See also: GRIPonMASH consortium website — https://griponmash.eu/